CLINICAL TRIAL: NCT04296435
Title: Observational Study About the Weekend Effect and Its Possible Influence on the Prognosis of Patients With Non-varicose Gastrointestinal Bleeding
Brief Title: The Weekend Effect and Its Possible Influence on the Prognosis of Patients With Non-varicose Upper Gastrointestinal Bleeding
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Other Study IDs: IIBSP-FIN-2018-50
Record Dates: First submitted 2020-03-03; First posted 2020-03-05 (Actual); Last update posted 2020-03-05 (Actual); Status verified 2020-03

CONDITIONS: Acute Upper Gastrointestinal Hemorrhage
Keywords: Weekend effect; non-varicose upper gastrointestinal bleeding

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The hypothesis is that the mortality of patients with non-varicose upper gastrointestinal bleeding after performing early gastroscopy who are admitted on weekends and night hours is higher than those admitted on weekdays or during daytime hours.

DETAILED DESCRIPTION:
The aim of the study is to evaluate the impact of the schedule (day or night) and the day of admission (working or weekend / night) on the mortality of patients with non-varicose upper gastrointestinal bleeding after performing an early gastroscopy.

A retrospective observational study will be carried out in patients admitted to the bleeding unit of the Santa Creu I Sant Pau Hospital, where we observed hospital mortality and 30 days after performing an early gastroscopy, the duration of admission, signs of hemorrhagic activity in a period of less than 12 h. After early gastroscopy and types of endoscopic treatments, data will be collected by reviewing medical records.

The number of patients expected to be included in this study is 1320 patients. Patients will be included the day they enter the bleeding unit for an early gastroscopy.

ELIGIBILITY:
Inclusion criteria:

* Patients older than 18 years.
* Patients admitted to the Bleeding Unit with a diagnosis of upper gastrointestinal bleeding.
* Patients who have undergone an early endoscopy to determine the source of bleeding.
* In case of readmissions during the study period, we consider only the admission closest to his death or discharge.

Exclusion criteria:

* Patients diagnosed with gastrointestinal bleeding varicose.
* Patients who present with gastrointestinal bleeding and did not perform early gastroscopy (during the first 24 hours)
* Patients admitted for different medical conditions, who developed upper gastrointestinal bleeding during the course of hospital stay.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with non-varicose upper gastrointestinal bleeding and admitted to the Bleeding Unit of the Santa Creu and Sant Pau hospital during 2017 and 2018 to perform an early gastroscopy. In addition, patients must meet the following inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 1320 (Estimated)
Dates: Start 2019-10-28 (Actual); Primary Completion 2021-10-28 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Mortality | During the years 2017 and 2018
  In-hospital mortality and at 30 days after early gastroscopy will be assessed through clinical history observation, within the study period

SECONDARY OUTCOMES:
Entry Duration | During the years 2017 and 2018
  The time between admission and discharge
Signs of bleeding activity in a period of less than 12 h. post gastroscopy early. | During the years 2017 and 2018
  It will be evaluated using the Rockall scale
Type of endoscopic treatments | During the years 2017 and 2018
  Hemostasis can be performed by applying different techniques or a combination of them

CONTACTS AND LOCATIONS:
Overall Officials: Luzdivina Perez Garcia, Principal Investigator — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Spain